CLINICAL TRIAL: NCT01210495
Title: A MULTICENTER, GLOBAL, RANDOMIZED, DOUBLE-BLIND STUDY OF AXITINIB PLUS BEST SUPPORTIVE CARE VERSUS PLACEBO PLUS BEST SUPPORTIVE CARE IN PATIENTS WITH ADVANCED HEPATOCELLULAR CARCINOMA FOLLOWING FAILURE OF ONE PRIOR ANTIANGIOGENIC THERAPY
Brief Title: Axitinib For The Treatment Of Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4061058; 2010-021590-37 (EudraCT Number)
Record Dates: First submitted 2010-09-22; First posted 2010-09-28 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Axitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Participants in this group received axitinib + best supportive care. Participants with Child-Pugh Class A disease (score 5 or 6) were enrolled into the randomized portion at a starting axitinib dose of 5 mg BID orally. Participants with Child-Pugh Class B disease (score 7) were to begin enrollment into the randomized portion of the study following determination of the recommended axitinib starting dose in the non-randomized portion. Study treatment was administered in cycles of 4 weeks in duration
  Interventions: Drug: Axitinib (AG-013736); Other: Best Supportive Care
- B (Placebo Comparator): Participants in this group received placebo + best supportive care. Treatment was administered in cycles of 4 weeks in duration. The starting dose of placebo for participants with Child Pugh Class A disease (score 5 or 6) was chosen as 5 mg BID. Participants with Child-Pugh Class B, score 7 received placebo that was determined from the non-randomized portion of the study until the recommended starting dose was determined, participants with Child-Pugh Class B, score 7, were not permitted to enter the randomized portion of the study
  Interventions: Drug: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: Axitinib (AG-013736) — Axitinib [tablet, 1 mg, 5 mg] will be given twice daily [BID] with continuous dosing; duration is approximately 3-6 months; starting dose is 5 mg BID
  Arms: A
Other: Best Supportive Care — BSC may include medications and supportive measures deemed necessary to palliate disease related symptoms and improve quality of life.
  Arms: A
Drug: Placebo — Placebo [tablet, 1 mg, 5 mg] will be given twice daily [BID] with continuous dosing; duration is approximately 3-6 months; starting dose is 5 mg BID
  Arms: B
Other: Best Supportive Care — BSC may include medications and supportive measures deemed necessary to palliate disease related symptoms and improve quality of life.
  Arms: B

SUMMARY:
The study is designed to demonstrate that axitinib plus best supportive care is superior to placebo plus best supportive care in prolonging survival in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic HCC
* Failure of one prior antiangiogenic therapy including sorafenib, bevacizumab and brivanib.
* Child-Pugh Class A or B (score 7 only) disease.

Exclusion Criteria:

* Prior treatment of advanced HCC with more than one prior first-line systemic therapy.
* Any prior local therapy within 2 weeks of starting the study treatment.
* Presence of hepatic encephalopathy and/or clinically relevant ascites.
* Presence of main portal vein invasion by HCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2010-12-06 (Actual); Primary Completion 2014-03-03 (Actual); Study Completion 2016-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (76):
- United States (12):
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - UCSD Medical Center- La Jolla, La Jolla, California
  - Moores UCSD Cancer Center, La Jolla, California
  - University of California Irvine Medical Center, Orange, California
  - UCSD Medical Center- Hillcrest, San Diego, California
  - Florida Hospital Transplant Center, Liver Unit, Orlando, Florida
  - Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - CHC Clinique Saint-Joseph, Liège
- China (7):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Jiang Su Cancer Hospital, Nanjing, Jiangsu
  - Sir Run Run Shaw Hospital of College of Medicine of Zhejiang University, Hangzhou, Zhejiang
  - The PLA 307 Hospital, Beijing
  - Zhongshan Hospital Fudan University, Shanghai
- France (11):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Hopital Saint André, Bordeaux
  - CHU Cote de Nacre, Caen
  - Bichat-Beaujon Service Inter Hospitalier De Cancerologie, Clichy
  - Hopital De La Croix-Rousse, Lyon
  - UPCET-CIC Timone, Marseille
  - CHRU Montpellier-Hopital Saint Eloi - Departement Oncologie Medicale, Montpellier
  - Hôpital L'Archet Ii, Nice
  - Hôpital Saint Antoine, Paris
  - Centre Eugène Marquis, Rennes
  - CHRU de Purpan., Toulouse
- Germany (3):
  - Medizinische Klinik mit Schwerpunkt, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinikum der Ludwig-Maximilians-Universitaet , Campus Grosshadern, München
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, N.T., HONG KONG
  - Queen Mary Hospital, Hong Kong
- Hungary (2):
  - Semmelweis Egyetem I.sz. Belgyógyászati Klinika, Budapest
  - Szegedi Tudományegyetem Onkoterápiás Klinika, Szeged
- Italy (8):
  - Istituto di Ematologia ed Oncologia Medica, Lorenzo ed Ariosto Seragnoli,, Bologna
  - Policlinico S.Orsola-Malpighi Dipartimento di Ematologia e Scienze Oncologiche "L. E A. Seragnoli", Bologna
  - Ospedale Versilia,Oncologia Medica, Lido Di Camaiore (LU)
  - Istituto Scientifico Romagnolo per lo Studio e la cura dei Tumori IRST, Meldola (FC)
  - Unita Operativa Oncologia Medica IRCCS Fondazione Salvatore Maugeri, Pavia
  - Policlinico Universitario Agostino Gemelli, Roma
  - Unità Operativa Oncologica Medica, Roma
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria aile Scotte, Siena
- Japan (9):
  - Aichi Cancer Center Central Hospital, Diagnostic and Interventional Radiology, Nagoya, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - Gifu Municipal Hospital, Gifu, Gifu
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kinki University Hospital, Ōsaka-sayama, Osaka
  - Shizuoka Cancer Center, Suntou-gun, Shizuoka
  - Sasaki Foundation Kyoundo Hospital, Chiyoda-Ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-Ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta Banska Bystrica, Banská Bystrica
  - Narodny onkologicky ustav, Bratislava
  - POKO Poprad s.r.o., Poprad
  - Nemocnica Poprad, a.s., Poprad
- South Korea (3):
  - National Cancer Center/ Center for Liver Cancer, Goyang-si
  - Samsung Medical Center, Division of Hematology-Oncology, Department of Medicine, Seoul
  - Asan Medical Center, Division of Oncology, Department of Internal Medicine, Seoul
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi-Mei Medical Center LiouYing, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan District
- United Kingdom (6):
  - The Christie NHS Foundation Trust, Withington, Manchester
  - Clatterbridge Centre for Oncology NHS Foundation Trust, Liverpool
  - Royal Liverpool and Broadgreen University Hospital, Liverpool
  - Royal Free Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kang YK, Yau T, Park JW, Lim HY, Lee TY, Obi S, Chan SL, Qin S, Kim RD, Casey M, Chen C, Bhattacharyya H, Williams JA, Valota O, Chakrabarti D, Kudo M. Randomized phase II study of axitinib versus placebo plus best supportive care in second-line treatment of advanced hepatocellular carcinoma. Ann Oncol. 2015 Dec;26(12):2457-63. doi: 10.1093/annonc/mdv388. Epub 2015 Sep 18. PMID 26386123
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061058&StudyName=Axitinib%20For%20The%20Treatment%20Of%20Advanced%20Hepatocellular%20Carcinoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 224 participants were enrolled in the study. Randomized portion enrolled 202 participants in 2 arms (134 in axitinib, 68 in placebo) in 70 centers (13 countries). Non-randomized portion enrolled 22 participants in 2 cohorts (15 in Child-Pugh Class A, 7 in Child-Pugh Class B score 7) according to Child-Pugh score in 13 centers (4 countries).
Pre-assignment Details: Participants with Child-Pugh Class A (score 5 or 6) could have been enrolled into either non-randomized or to randomized portion. Participants with Child-Pugh Class B (score 7) were initially enrolled into non-randomized portion but following determination of recommended axitinib starting dose they could have been enrolled in randomized portion.
Groups:
- Child-Pugh Class A: Participants with Child-Pugh Class A disease (score 5 or 6) were enrolled into the non-randomized portion at selected sites only at a starting axitinib dose of 5 milligrams (mg) twice daily (BID).
- Child-Pugh Class B: Participants with Child-Pugh Class B disease (score 7) at selected sites were initially enrolled only into the non-randomized portion of this study to determine the recommended starting dose of axitinib for this population. The initial starting dose for this group was 2 mg BID.
- Axitinib: Participants in this group received axitinib + best supportive care. Participants with Child-Pugh Class A disease (score 5 or 6) were enrolled into the randomized portion at a starting axitinib dose of 5 mg BID orally. Participants with Child-Pugh Class B disease (score 7) were to begin enrollment into the randomized portion of the study following determination of the recommended axitinib starting dose in the non-randomized portion. Study treatment was administered in cycles of 4 weeks in duration (up to a maximum of 55 cycles).
- Placebo: Participants in this group received placebo + best supportive care. Treatment was administered in cycles of 4 weeks in duration (up to a maximum of 55 cycles). The starting dose of placebo for participants with Child Pugh Class A disease (score 5 or 6) was chosen as 5 mg BID. Participants with Child-Pugh Class B, score 7 received placebo that was determined from the non-randomized portion of the study until the recommended starting dose was determined, participants with Child-Pugh Class B, score 7, were not permitted to enter the randomized portion of the study.
Period: Overall Study
Arm/Group | Child-Pugh Class A | Child-Pugh Class B | Axitinib | Placebo
Started | 15 | 7 | 134 | 68
Completed | 0 | 0 | 0 | 0
Not Completed | 15 | 7 | 134 | 68
Not completed — Participant Refused Further Follow-Up | 1 | 0 | 11 | 2
Not completed — Death | 14 | 7 | 112 | 54
Not completed — Study Terminated by Sponsor | 0 | 0 | 4 | 11
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Other unspecified | 0 | 0 | 6 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants, and participants were classified according to the randomized treatment arm regardless of what treatment, if any, was received.
Groups:
- Child-Pugh Class A: Participants with Child-Pugh Class A disease (score 5 or 6) were enrolled into the non-randomized portion at selected sites only at a starting axitinib dose of 5 mg BID.
- Axitinib: Participants in this group received axitinib + best supportive care. Participants with Child-Pugh Class A disease (score 5 or 6) were enrolled into the randomized portion at a starting axitinib dose of 5 mg BID orally. Participants with Child-Pugh Class B disease (score 7) were to begin enrollment into the randomized portion of the study following determination of the recommended axitinib starting dose in the non randomized portion. Study treatment was administered in cycles of 4 weeks in duration (up to a maximum of 55 cycles).
- Placebo: Participants in this group received placebo + best supportive care. Treatment was administered in cycles of 4 weeks in duration (up to a maximum of 55 cycles). The starting dose of placebo for participants with Child Pugh Class A disease (score 5 or 6) was chosen as 5 mg BID. Participants with Child-Pugh Class B, score 7 received placebo that was determined from the non-randomized portion of the study until the recommended starting dose was determined, participants with Child Pugh Class B, score 7, were not permitted to enter the randomized portion of the study.
- Total: Total of all reporting groups
Arm/Group | Child-Pugh Class A | Child-Pugh Class B | Axitinib | Placebo | Total
Number analyzed (Participants) | 15 | 7 | 134 | 68 | 224
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0
  18-44 years | 4 | 0 | 7 | 4 | 15
  45-64 years | 5 | 5 | 74 | 32 | 116
  >=65 years | 6 | 2 | 53 | 32 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 24 | 12 | 41
  Male | 12 | 5 | 110 | 56 | 183

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) - Stratified Analysis, Randomized Portion
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. OS (in months) was calculated as (date of death - first randomization date +1)/30.4. For participants still alive at the time of the analysis, the OS time was censored on the last date they were known to be alive. All participants were followed up for survival at least every 3 months after discontinuing study treatment until at least two years after randomization of the last participant.
Time Frame: From randomization until at least two years after the last participant has been randomized (up to 6 years)
Population: FAS included all randomized participants, and participants were classified according to the randomized treatment arm regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
months | 12.7 [10.2 to 14.9] | 9.7 [5.9 to 11.8]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; The study was designed to test the null hypothesis that the true median OS was 5 months vs. the alternative hypothesis that the true median OS was at least 8.3 months (i.e., 66 percent [%] improvement in median OS); Test type: Superiority or Other; p = 0.2872, Log Rank — For the overall stratified analysis the p-value is from a 1-sided log-rank test of treatment stratified by tumor invasion and geographic region; Hazard Ratio (HR) = 0.907, 95% CI 2-sided [0.646 to 1.274] — Assuming proportional hazards, a hazard ratio less than (<) 1 indicated reduction in hazard rate to favor Axitinib; hazard ratio greater than (>) 1 indicated reduction to favor Placebo

2. Secondary Outcome: Progression-Free Survival (PFS) - Stratified Analysis, Randomized Portion
Description: PFS was defined as time from randomization to first documented objective tumor progression or to death due to any cause, whichever occurred first. PFS (in months) was calculated as (first event date - first randomization date +1)/30.4. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was death). As per response evaluation criteria in solid tumors (RECIST) 1.1, progression was defined as greater than or equal to (>=) 20% increase in sum of longest dimensions of target lesions or appearance of one or more new target lesions and unequivocal progression of existing non-target lesions, or appearance of 1 new non-target lesions. Participants discontinuing study treatment without documented evidence of PD were to be followed up at least every 8 weeks after discontinuing study treatment until disease progression, or initiation of another anticancer treatment.
Time Frame: Every 8 weeks until disease progression/death or start of new treatment or until at least two years after the last participant has been randomized, whatever occurs first
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
months | 3.6 [2.3 to 4.6] | 1.9 [1.9 to 3.5]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Test type: Superiority or Other; p = 0.0039, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.618, 95% CI 2-sided [0.438 to 0.871] — Assuming proportional hazards, a hazard ratio <1 indicated a reduction in hazard rate in favor of Axitinib; a hazard ratio >1 indicated a reduction in favor of Placebo

3. Secondary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response by Stratified Analysis, Randomized Portion
Description: ORR was defined as the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR) according to the RECIST 1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must decrease to normal (short axis <10 millimetres [mm]). PR was defined as a 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Every 8 weeks until at least two years after the last participant has been randomized
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
percentage of participants | 9.7 [5.3 to 16.0] | 2.9 [0.4 to 10.2]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Test type: Superiority or Other; p = 0.0914, Cochran-Mantel-Haenszel — ORR for the 2 treatment arms was compared with a significance level of 0.025 using Cochran-Mantel-Haenszel (CMH) test for stratified analyses; Risk Ratio (RR) = 3.172, 95% CI 2-sided [0.759 to 13.265] — Risk ratio and confidence interval (CI) were based on the Mantel-Haenszel estimator; risk ratio was adjusted for geographical region and vascular invasion and extra hepatic spread

4. Secondary Outcome: Time to Tumor Progression (TTP) - Stratified Analysis, Randomized Portion
Description: TTP was defined as the time from randomization to first documentation of objective tumor progression. If tumor progression data included more than 1 date, the first date was used. TTP (in months) was calculated as (first event date - first randomization date +1)/30.4.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
months | 3.7 [2.8 to 5.6] | 1.9 [1.9 to 3.6]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Test type: Superiority or Other; p = 0.006, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.621, 95% CI 2-sided [0.434 to 0.889] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Duration of Response (DR) by Unstratified Analysis, Randomized Portion
Description: DR was defined as the time from the first documentation of objective tumor response (CR or PR) that was subsequently confirmed to the first documentation of PD or to death due to any cause, whichever occurs first. If tumor progression data included more than 1 date, the first date was to be used. DR (in months) was to be calculated as (the end date for DR - first CR or PR that was subsequently confirmed +1)/30.4.
Time Frame: From objective response to date of progression or death
Population: FAS included all randomized participants, and participants were classified according to the randomized treatment arm regardless of what treatment, if any, was received. DR was calculated for the subgroup of FAS participants with objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 13 | 2
months | 6.4 [3.7 to 9.3] | NA [NA to NA] — Not reached

6. Secondary Outcome: Percentage of Participants With Overall Clinical Benefit Response (CBR) - Stratified Analysis, Randomized Portion
Description: CBR was defined as the percentage of participants with confirmed CR or confirmed PR or a best response of stable disease >=8 weeks according to RECIST 1.1 criteria, relative to all randomized participants who had baseline measurable disease. Confirmed responses were defined as those that persisted on repeat imaging study >=4 weeks after the initial documentation of response. Participants who did not have on study radiographic tumor re-evaluation or who died, progressed, or dropped out for any reason prior to reaching a CR, PR, or stable disease were counted as non-responders in the assessment of CBR. A participant who initially met the criteria for a PR and then subsequently became a confirmed CR was to be assigned a best response of CR.
Time Frame: From Baseline up to end of treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
percentage of participants | 31.3 [23.6 to 39.9] | 11.8 [5.2 to 21.9]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Test type: Superiority or Other; p = 0.0025, Cochran-Mantel-Haenszel — For the overall stratified analysis the p-value is from Cochran-Mantel-Haenszel test of treatment stratified by geographical region and vascular invasion and extra hepatic spread; Risk Ratio (RR) = 2.650, 95% CI 2-sided [1.319 to 5.326] — Risk Ratio and CI based on the Mantel-Haenszel estimator; risk ratio was adjusted for geographical region and vascular invasion and extra hepatic spread

7. Secondary Outcome: Axitinib Steady-State Pharmacokinetic (PK) Parameter - Maximum Observed Plasma Concentration (Cmax), Non-Randomized Portion
Description: Axitinib samples were to be collected from all participants on Cycle 1 Day 15 at the following time points: pre-dose, 1, 2, 3, 4, 6 and 8 hours after axitinib dosing.
Time Frame: Cycle 1 Day 15
Population: The PK concentration set included all participants who were treated and had at least 1 measured concentration on at least 1 day of PK assessment. The PK parameter analysis set included all participants treated who had at least 1 estimated PK parameter of primary interest.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 12 | 7
nanograms per milliliter (ng/mL) | 35.74 [21.84 to 58.50] | 21.16 [11.10 to 40.33]

8. Secondary Outcome: Axitinib Steady-State PK Parameter - Area Under the Plasma Concentration Versus Time Curve From 0 to 24 Hour (AUC0-24), Non-Randomized Portion
Description: Axitinib samples were to be collected from all participants on Cycle 1 Day 15 at the following time points: pre-dose, 1, 2, 3, 4, 6 and 8 hours after axitinib dosing. In the below table, 4 participants in Child-Pugh A and 1 participant in Child-Pugh B were not reported due to nonestimable half-life.
Time Frame: Cycle 1 Day 15
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 8 | 6
nanograms*hour per milliliter (ng*hr/mL) | 310.76 [175.02 to 551.75] | 316.20 [162.96 to 613.55]

9. Secondary Outcome: Axitinib Steady-State Pharmacokinetic Parameter - Time to First Occurrence of Cmax (Tmax), Non-Randomized Portion
Description: as for outcome 7
Time Frame: Cycle 1 Day 15
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 12 | 7
hours | 2.50 [0.00 to 7.98] | 1.05 [0.00 to 4.00]

10. Secondary Outcome: Axitinib Steady-State Pharmacokinetic Parameter - Apparent Oral Clearance (CL/F), Non-Randomized Portion
Description: as for outcome 8
Time Frame: Cycle 1 Day 15
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: liters per hour (L/hr)
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 8 | 6
liters per hour (L/hr) | 32.18 [18.12 to 57.13] | 12.65 [6.52 to 24.55]

11. Secondary Outcome: Axitinib Steady-State Pharmacokinetic Parameter - Terminal Plasma Elimination Half-Life (t1/2), Non-Randomized Portion
Description: as for outcome 8
Time Frame: Cycle 1 Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 8 | 6
hours | 4.12 (3.55) [18.12 to 57.13] | 4.79 (2.42) [6.52 to 24.55]

12. Secondary Outcome: Axitinib Steady-State Pharmacokinetic Parameter - Apparent Oral Volume of Distribution of the Drug During the Elimination Phase (Vz/F), Non-Randomized Portion
Description: Axitinib samples were to be collected from all participants on Cycle 1 Day 15 at the following time points: pre-dose, 1, 2, 3, 4, 6 and 8 hours after axitinib dosing. The PK parameter, Vz/F has been presented in this outcome measure. In the below table, 4 participants in Child-Pugh A and 1 participant in Child-Pugh B were not reported due to nonestimable half-life.
Time Frame: Cycle 1 Day 15
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: liters
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 8 | 6
liters | 150.01 (3.55) [94.67 to 237.68] | 81.16 (2.42) [47.70 to 138.08]

13. Secondary Outcome: Concentration of Soluble Proteins at Baseline in Randomized Portion
Description: Plasma soluble proteins interleukin-6 (IL-6), E-Selectin, interleukin-8 (IL-8), hepatocyte growth factor (HGF), matrix metalloproteinase-2 (MMP-2), stem cell factor (SCF), angiopoietin-2 (Ang-2), vascular endothelial growth factor-A (VEGF-A), vascular endothelial growth factor-C (VEGF-C), soluble vascular endothelial growth factor receptor 2 (sVEGFR2), soluble vascular endothelial growth factor receptor 3 (sVEGFR3), stromal cell-derived factor-1 (SDF1), neutrophil gelatinase-associated lipocalin (NGAL), migration inhibitory factor (MIF), c-MET, regulated upon activation normal T cell expressed and presumably secreted (RANTES), and monocyte chemotactic protein-3 (MCP-3) were only measured in randomized participants.
Time Frame: Baseline
Population: The soluble protein analysis set included all participants in the safety analysis set who had a Baseline soluble protein assessment. Safety analysis population included all randomized participants who received at least 1 dose of study drug with treatment assignments designated according to actual study treatment received.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 120 | 61
picograms per milliliter (pg/mL)
  IL-6 | 50.67 (102.86) | 50.72 (106.74)
  E-Selectin | 52313.94 (32603.18) | 55430.76 (26723.43)
  IL-8 | 33.35 (47.72) | 27.23 (44.46)
  HGF | 478.84 (712.43) | 406.06 (376.04)
  MMP-2 | 355715.66 (137663.04) | 350979.72 (146323.29)
  SCF | 1352.75 (1534.41) | 1439.71 (2260.89)
  Ang-2 | 662.40 (623.87) | 577.82 (354.42)
  VEGF-A | 102.56 (128.09) | 173.59 (472.19)
  VEGF-C | NA (NA) — Not available as the % < LLQ (lower limit of quantification) was greater than 75%. | NA (NA) — Not available as the % < LLQ was greater than 75%.
  sVEGFR2 | 17675.76 (7218.95) | 18273.65 (6836.16)
  sVEGFR3 | 287429.28 (117583.24) | 290338.69 (97830.36)
  SDF1 | 1190.08 (823.03) | 1150.10 (681.04)
  NGAL | 134861.80 (152492.96) | 141383.00 (121747.35)
  MIF | 33057.15 (28256.00) | 32302.99 (21485.01)
  c-MET ELISA | 1664.96 (834.36) | 1641.08 (704.38)
  RANTES | 26412.12 (38682.81) | 26917.76 (27094.12)
  MCP-3 | NA (NA) — Not available as the % < LLQ was greater than 75%. | NA (NA) — Not available as the % < LLQ was greater than 75%.

14. Secondary Outcome: Percentage of Participants With Specific Micro-Ribonucleic Acid (miRNA) Transcript Present in Circulation in Randomized Portion
Description: A 5 millilitres (mL) whole blood sample was collected from all randomized participants to evaluate the miRNA transcripts.
Time Frame: Baseline
Population: The miRNA analysis set included all participants in the safety analysis set who had a baseline miRNA assessment. Safety analysis population included all randomized participants who received at least 1 dose of study drug with treatment assignments designated according to actual study treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 111 | 59
percentage of participants
  hsa-let-7a-5p | 100.0 | 100.0
  hsa-let-7b-5p | 100.0 | 100.0
  hsa-let-7c | 100.0 | 100.0
  hsa-let-7d-5p | 100.0 | 100.0
  hsa-let-7f-5p | 100.0 | 100.0
  hsa-let-7g-5p | 100.0 | 100.0
  hsa-let-7i-5p | 100.0 | 100.0
  hsa-miR-103a-3p | 100.0 | 100.0
  hsa-miR-106b-5p | 100.0 | 100.0
  hsa-miR-107 | 100.0 | 100.0
  hsa-miR-1202 | 100.0 | 100.0
  hsa-miR-1207-5p | 100.0 | 100.0
  hsa-miR-1225-5p | 100.0 | 100.0
  hsa-miR-1234-5p | 100.0 | 100.0
  hsa-miR-1246 | 100.0 | 100.0
  hsa-miR-125b-5p | 100.0 | 100.0
  hsa-miR-126-3p | 100.0 | 100.0
  hsa-miR-1260a | 100.0 | 100.0
  hsa-miR-1260b | 100.0 | 100.0
  hsa-miR-1268a | 100.0 | 100.0
  hsa-miR-1273g-3p | 100.0 | 100.0
  hsa-miR-1275 | 100.0 | 100.0
  hsa-miR-128 | 100.0 | 100.0
  hsa-miR-130a-3p | 100.0 | 100.0
  hsa-miR-130b-3p | 100.0 | 100.0
  hsa-miR-140-3p | 100.0 | 100.0
  hsa-miR-142-3p | 100.0 | 100.0
  hsa-miR-145-5p | 100.0 | 100.0
  hsa-miR-148a-3p | 100.0 | 100.0
  hsa-miR-148b-3p | 100.0 | 100.0
  hsa-miR-150-5p | 100.0 | 100.0
  hsa-miR-151a-3p | 100.0 | 100.0
  hsa-miR-151a-5p | 100.0 | 100.0
  hsa-miR-151b | 100.0 | 100.0
  hsa-miR-1587 | 100.0 | 100.0
  hsa-miR-15a-5p | 100.0 | 100.0
  hsa-miR-15b-5p | 100.0 | 100.0
  hsa-miR-16-5p | 100.0 | 100.0
  hsa-miR-17-5p | 100.0 | 100.0
  hsa-miR-181a-5p | 100.0 | 100.0
  hsa-miR-182-5p | 100.0 | 100.0
  hsa-miR-183-5p | 100.0 | 100.0
  hsa-miR-185-5p | 100.0 | 100.0
  hsa-miR-186-5p | 100.0 | 100.0
  hsa-miR-191-5p | 100.0 | 100.0
  hsa-miR-1914-3p | 100.0 | 100.0
  hsa-miR-1915-3p | 100.0 | 100.0
  hsa-miR-192-5p | 100.0 | 100.0
  hsa-miR-194-5p | 100.0 | 100.0
  hsa-miR-197-3p | 100.0 | 100.0
  hsa-miR-197-5p | 100.0 | 100.0
  hsa-miR-19a-3p | 100.0 | 100.0
  hsa-miR-19b-3p | 100.0 | 100.0
  hsa-miR-20a-5p | 100.0 | 100.0
  hsa-miR-20b-5p | 100.0 | 100.0
  hsa-miR-21-5p | 100.0 | 100.0
  hsa-miR-210 | 100.0 | 100.0
  hsa-miR-215 | 100.0 | 100.0
  hsa-miR-22-3p | 100.0 | 100.0
  hsa-miR-222-3p | 100.0 | 100.0
  hsa-miR-223-3p | 100.0 | 100.0
  hsa-miR-23a-3p | 100.0 | 100.0
  hsa-miR-23b-3p | 100.0 | 100.0
  hsa-miR-24-3p | 100.0 | 100.0
  hsa-miR-25-3p | 100.0 | 100.0
  hsa-miR-26a-5p | 100.0 | 100.0
  hsa-miR-26b-5p | 100.0 | 100.0
  hsa-miR-2861 | 100.0 | 100.0
  hsa-miR-29a-3p | 100.0 | 100.0
  hsa-miR-29b-3p | 100.0 | 100.0
  hsa-miR-29c-3p | 100.0 | 100.0
  hsa-miR-29c-5p | 100.0 | 100.0
  hsa-miR-30b-5p | 100.0 | 100.0
  hsa-miR-30c-5p | 100.0 | 100.0
  hsa-miR-30d-5p | 100.0 | 100.0
  hsa-miR-30e-5p | 100.0 | 100.0
  hsa-miR-3135b | 100.0 | 100.0
  hsa-miR-3162-5p | 100.0 | 100.0
  hsa-miR-3180-3p | 100.0 | 100.0
  hsa-miR-3195 | 100.0 | 100.0
  hsa-miR-320a | 100.0 | 100.0
  hsa-miR-320b | 100.0 | 100.0
  hsa-miR-320c | 100.0 | 100.0
  hsa-miR-320d | 100.0 | 100.0
  hsa-miR-320e | 100.0 | 100.0
  hsa-miR-324-3p | 100.0 | 100.0
  hsa-miR-324-5p | 100.0 | 100.0
  hsa-miR-331-3p | 100.0 | 100.0
  hsa-miR-339-5p | 100.0 | 100.0
  hsa-miR-342-3p | 100.0 | 100.0
  hsa-miR-361-3p | 100.0 | 100.0
  hsa-miR-361-5p | 100.0 | 100.0
  hsa-miR-362-5p | 100.0 | 100.0
  hsa-miR-363-3p | 100.0 | 100.0
  hsa-miR-3651 | 100.0 | 100.0
  hsa-miR-3656 | 100.0 | 100.0
  hsa-miR-365a-3p | 100.0 | 100.0
  hsa-miR-3665 | 100.0 | 100.0
  hsa-miR-3676-5p | 100.0 | 100.0
  hsa-miR-374b-5p | 100.0 | 100.0
  hsa-miR-378a-3p | 100.0 | 100.0
  hsa-miR-378i | 100.0 | 100.0
  hsa-miR-3940-5p | 100.0 | 100.0
  hsa-miR-3960 | 100.0 | 100.0
  hsa-miR-423-3p | 100.0 | 100.0
  hsa-miR-425-5p | 100.0 | 100.0
  hsa-miR-4281 | 100.0 | 100.0
  hsa-miR-4284 | 100.0 | 100.0
  hsa-miR-4286 | 100.0 | 100.0
  hsa-miR-4299 | 100.0 | 100.0
  hsa-miR-4306 | 100.0 | 100.0
  hsa-miR-4318 | 100.0 | 100.0
  hsa-miR-4323 | 100.0 | 100.0
  hsa-miR-4428 | 100.0 | 100.0
  hsa-miR-4442 | 100.0 | 100.0
  hsa-miR-4443 | 100.0 | 100.0
  hsa-miR-4454 | 100.0 | 100.0
  hsa-miR-4459 | 100.0 | 100.0
  hsa-miR-4466 | 100.0 | 100.0
  hsa-miR-4497 | 100.0 | 100.0
  hsa-miR-4505 | 100.0 | 100.0
  hsa-miR-4507 | 100.0 | 100.0
  hsa-miR-4516 | 100.0 | 100.0
  hsa-miR-451a | 100.0 | 100.0
  hsa-miR-4530 | 100.0 | 100.0
  hsa-miR-4687-3p | 100.0 | 100.0
  hsa-miR-4713-3p | 100.0 | 100.0
  hsa-miR-4721 | 100.0 | 100.0
  hsa-miR-4728-5p | 100.0 | 100.0
  hsa-miR-4732-3p | 100.0 | 100.0
  hsa-miR-4739 | 100.0 | 100.0
  hsa-miR-4763-3p | 100.0 | 100.0
  hsa-miR-4787-5p | 100.0 | 100.0
  hsa-miR-4788 | 100.0 | 100.0
  hsa-miR-484 | 100.0 | 100.0
  hsa-miR-486-5p | 100.0 | 100.0
  hsa-miR-494 | 100.0 | 100.0
  hsa-miR-5001-5p | 100.0 | 100.0
  hsa-miR-500a-3p | 100.0 | 100.0
  hsa-miR-500a-5p | 100.0 | 100.0
  hsa-miR-501-3p | 100.0 | 100.0
  hsa-miR-501-5p | 100.0 | 100.0
  hsa-miR-502-3p | 100.0 | 100.0
  hsa-miR-505-5p | 100.0 | 100.0
  hsa-miR-5100 | 100.0 | 100.0
  hsa-miR-532-3p | 100.0 | 100.0
  hsa-miR-532-5p | 100.0 | 100.0
  hsa-miR-550a-3-5p | 100.0 | 100.0
  hsa-miR-550a-3p | 100.0 | 100.0
  hsa-miR-5739 | 100.0 | 100.0
  hsa-miR-574-3p | 100.0 | 100.0
  hsa-miR-574-5p | 100.0 | 100.0
  hsa-miR-5787 | 100.0 | 100.0
  hsa-miR-584-5p | 100.0 | 100.0
  hsa-miR-6085 | 100.0 | 100.0
  hsa-miR-6087 | 100.0 | 100.0
  hsa-miR-6088 | 100.0 | 100.0
  hsa-miR-6089 | 100.0 | 100.0
  hsa-miR-6090 | 100.0 | 100.0
  hsa-miR-6125 | 100.0 | 100.0
  hsa-miR-6127 | 100.0 | 100.0
  hsa-miR-625-5p | 100.0 | 100.0
  hsa-miR-638 | 100.0 | 100.0
  hsa-miR-642a-3p | 100.0 | 100.0
  hsa-miR-642b-3p | 100.0 | 100.0
  hsa-miR-652-3p | 100.0 | 100.0
  hsa-miR-660-5p | 100.0 | 100.0
  hsa-miR-664a-3p | 100.0 | 100.0
  hsa-miR-664b-3p | 100.0 | 100.0
  hsa-miR-6717-5p | 100.0 | 100.0
  hsa-miR-6724-5p | 100.0 | 100.0
  hsa-miR-7-5p | 100.0 | 100.0
  hsa-miR-762 | 100.0 | 100.0
  hsa-miR-766-3p | 100.0 | 100.0
  hsa-miR-92a-3p | 100.0 | 100.0
  hsa-miR-93-3p | 100.0 | 100.0
  hsa-miR-93-5p | 100.0 | 100.0
  hsa-miR-937-5p | 100.0 | 100.0
  hsa-miR-940 | 100.0 | 100.0
  hsa-miR-1228-3p | 99.1 | 100.0
  hsa-miR-1268b | 99.1 | 100.0
  hsa-miR-142-5p | 100.0 | 98.3
  hsa-miR-27a-3p | 99.1 | 100.0
  hsa-miR-296-5p | 99.1 | 100.0
  hsa-miR-3196 | 99.1 | 100.0
  hsa-miR-3198 | 99.1 | 100.0
  hsa-miR-342-5p | 100.0 | 98.3
  hsa-miR-3653 | 100.0 | 98.3
  hsa-miR-4465 | 99.1 | 100.0
  hsa-miR-4515 | 99.1 | 100.0
  hsa-miR-4653-3p | 99.1 | 100.0
  hsa-miR-4665-3p | 99.1 | 100.0
  hsa-miR-4746-3p | 99.1 | 100.0
  hsa-miR-505-3p | 100.0 | 98.3
  hsa-miR-6073 | 99.1 | 100.0
  hsa-miR-6126 | 99.1 | 100.0
  hsa-miR-6132 | 99.1 | 100.0
  hsa-miR-6165 | 99.1 | 100.0
  hsa-miR-744-5p | 100.0 | 98.3
  hsa-miR-874 | 99.1 | 100.0
  hsa-miR-942 | 100.0 | 98.3
  hsa-miR-96-5p | 99.1 | 100.0
  hsa-miR-1238-3p | 98.2 | 100.0
  hsa-miR-1285-3p | 99.1 | 98.3
  hsa-miR-1305 | 98.2 | 100.0
  hsa-miR-146a-5p | 98.2 | 100.0
  hsa-miR-15b-3p | 99.1 | 98.3
  hsa-miR-17-3p | 98.2 | 100.0
  hsa-miR-195-5p | 99.1 | 98.3
  hsa-miR-199a-5p | 99.1 | 98.3
  hsa-miR-28-5p | 99.1 | 98.3
  hsa-miR-30a-5p | 99.1 | 98.3
  hsa-miR-340-3p | 99.1 | 98.3
  hsa-miR-3679-5p | 99.1 | 98.3
  hsa-miR-374a-5p | 99.1 | 98.3
  hsa-miR-378a-5p | 99.1 | 98.3
  hsa-miR-4433-5p | 98.2 | 100.0
  hsa-miR-454-3p | 99.1 | 98.3
  hsa-miR-4685-5p | 99.1 | 98.3
  hsa-miR-575 | 98.2 | 100.0
  hsa-miR-6068 | 98.2 | 100.0
  hsa-miR-6124 | 98.2 | 100.0
  hsa-miR-6131 | 98.2 | 100.0
  hsa-miR-939-5p | 98.2 | 100.0
  hsa-miR-1234-3p | 99.1 | 96.6
  hsa-miR-1249 | 98.2 | 98.3
  hsa-miR-132-3p | 99.1 | 96.6
  hsa-miR-30e-3p | 98.2 | 98.3
  hsa-miR-326 | 99.1 | 96.6
  hsa-miR-374c-5p | 98.2 | 98.3
  hsa-miR-4270 | 97.3 | 100.0
  hsa-miR-4672 | 97.3 | 100.0
  hsa-miR-4741 | 98.2 | 98.3
  hsa-miR-6515-3p | 97.3 | 100.0
  hsa-miR-371b-5p | 97.3 | 98.3
  hsa-miR-4485 | 96.4 | 100.0
  hsa-miR-4513 | 98.2 | 96.6
  hsa-miR-454-5p | 98.2 | 96.6
  hsa-miR-4716-3p | 96.4 | 100.0
  hsa-miR-5006-5p | 97.3 | 98.3
  hsa-miR-6069 | 98.2 | 96.6
  hsa-miR-101-3p | 97.3 | 96.6
  hsa-miR-155-5p | 97.3 | 96.6
  hsa-miR-16-2-3p | 98.2 | 94.9
  hsa-miR-27b-3p | 98.2 | 94.9
  hsa-miR-328 | 98.2 | 94.9
  hsa-miR-4486 | 96.4 | 98.3
  hsa-miR-513a-5p | 96.4 | 98.3
  hsa-miR-92b-3p | 98.2 | 94.9
  hsa-miR-98-5p | 98.2 | 94.9
  hsa-miR-18b-5p | 96.4 | 96.6
  hsa-miR-191-3p | 97.3 | 94.9
  hsa-miR-3200-5p | 97.3 | 94.9
  hsa-miR-4313 | 97.3 | 94.9
  hsa-miR-4532 | 96.4 | 96.6
  hsa-miR-4787-3p | 97.3 | 94.9
  hsa-miR-513b | 95.5 | 98.3
  hsa-miR-550a-5p | 97.3 | 94.9
  hsa-miR-5581-5p | 94.6 | 100.0
  hsa-miR-629-3p | 97.3 | 94.9
  hsa-miR-629-5p | 94.6 | 100.0
  hsa-miR-7-1-3p | 98.2 | 93.2
  hsa-miR-125a-3p | 94.6 | 98.3
  hsa-miR-1281 | 97.3 | 93.2
  hsa-miR-140-5p | 95.5 | 96.6
  hsa-miR-144-5p | 96.4 | 94.9
  hsa-let-7b-3p | 96.4 | 93.2
  hsa-let-7f-1-3p | 95.5 | 94.9
  hsa-miR-125a-5p | 96.4 | 93.2
  hsa-miR-183-3p | 96.4 | 93.2
  hsa-miR-3162-3p | 97.3 | 91.5
  hsa-miR-33b-3p | 97.3 | 91.5
  hsa-miR-4669 | 94.6 | 96.6
  hsa-miR-502-5p | 96.4 | 93.2
  hsa-miR-1304-3p | 97.3 | 89.8
  hsa-miR-1306-5p | 95.5 | 93.2
  hsa-miR-221-3p | 93.7 | 96.6
  hsa-miR-4649-3p | 96.4 | 91.5
  hsa-miR-4690-5p | 94.6 | 94.9
  hsa-miR-627 | 95.5 | 93.2
  hsa-miR-99a-5p | 96.4 | 91.5
  hsa-miR-18a-5p | 94.6 | 93.2
  hsa-miR-211-3p | 94.6 | 93.2
  hsa-miR-4430 | 95.5 | 91.5
  hsa-miR-6508-5p | 95.5 | 91.5
  hsa-miR-933 | 95.5 | 91.5
  hsa-miR-339-3p | 94.6 | 91.5
  hsa-miR-624-5p | 95.5 | 89.8
  hsa-miR-425-3p | 95.5 | 88.1
  hsa-miR-5194 | 91.9 | 93.2
  hsa-miR-6511b-3p | 92.8 | 91.5
  hsa-let-7d-3p | 92.8 | 89.8
  hsa-miR-129-2-3p | 92.8 | 89.8
  hsa-miR-1825 | 92.8 | 89.8
  hsa-miR-362-3p | 93.7 | 88.1
  hsa-miR-665 | 91.0 | 93.2
  hsa-miR-149-5p | 92.8 | 88.1
  hsa-miR-3620-5p | 91.0 | 91.5
  hsa-miR-4478 | 90.1 | 91.5
  hsa-miR-4484 | 92.8 | 86.4
  hsa-miR-4656 | 90.1 | 91.5
  hsa-miR-602 | 91.9 | 88.1
  hsa-miR-1233-1-5p | 89.2 | 91.5
  hsa-miR-3125 | 89.2 | 91.5
  hsa-miR-4725-5p | 91.0 | 88.1
  hsa-miR-4732-5p | 91.0 | 88.1
  hsa-miR-146b-5p | 92.8 | 83.1
  hsa-miR-4659a-3p | 91.0 | 86.4
  hsa-miR-6510-5p | 88.3 | 91.5
  hsa-miR-1225-3p | 91.0 | 84.7
  hsa-miR-1539 | 90.1 | 86.4
  hsa-miR-188-5p | 88.3 | 89.8
  hsa-miR-4758-3p | 91.0 | 84.7
  hsa-miR-550b-2-5p | 91.9 | 83.1
  hsa-miR-144-3p | 89.2 | 86.4
  hsa-miR-4310 | 89.2 | 84.7
  hsa-miR-4749-3p | 89.2 | 84.7
  hsa-miR-1229-5p | 87.4 | 86.4
  hsa-miR-1288 | 86.5 | 88.1
  hsa-miR-3156-5p | 84.7 | 91.5
  hsa-miR-2116-3p | 89.2 | 81.4
  hsa-miR-4664-3p | 87.4 | 84.7
  hsa-miR-23c | 87.4 | 83.1
  hsa-miR-3652 | 85.6 | 86.4
  hsa-miR-424-5p | 88.3 | 81.4
  hsa-miR-4745-5p | 85.6 | 86.4
  hsa-miR-1973 | 83.8 | 88.1
  hsa-miR-4291 | 84.7 | 86.4
  hsa-miR-3200-3p | 86.5 | 81.4
  hsa-miR-4436b-5p | 84.7 | 84.7
  hsa-miR-6512-5p | 82.9 | 88.1
  hsa-miR-3613-3p | 86.5 | 78.0
  hsa-miR-4793-5p | 81.1 | 88.1
  hsa-miR-628-3p | 83.8 | 83.1
  hsa-miR-1181 | 82.9 | 83.1
  hsa-miR-3646 | 82.0 | 84.7
  hsa-miR-4317 | 82.9 | 83.1
  hsa-miR-5684 | 83.8 | 81.4
  hsa-miR-1227-5p | 81.1 | 84.7
  hsa-miR-3180-5p | 84.7 | 78.0
  hsa-miR-4665-5p | 82.9 | 81.4
  hsa-miR-129-1-3p | 82.0 | 81.4
  hsa-miR-4652-3p | 82.9 | 79.7
  hsa-miR-500b | 82.0 | 79.7
  hsa-miR-181b-5p | 83.8 | 74.6
  hsa-miR-3676-3p | 82.9 | 76.3
  hsa-miR-671-5p | 77.5 | 86.4
  hsa-miR-1185-1-3p | 78.4 | 83.1
  hsa-miR-378d | 78.4 | 83.1
  hsa-miR-1271-5p | 81.1 | 76.3
  hsa-miR-4433-3p | 78.4 | 81.4
  hsa-miR-564 | 81.1 | 76.3
  hsa-miR-6723-5p | 81.1 | 76.3
  hsa-miR-100-5p | 82.9 | 71.2
  hsa-miR-135a-3p | 77.5 | 81.4
  hsa-miR-181a-2-3p | 80.2 | 76.3
  hsa-miR-4666b | 78.4 | 79.7
  hsa-miR-98-3p | 79.3 | 76.3
  hsa-miR-3940-3p | 77.5 | 74.6
  hsa-miR-513c-5p | 74.8 | 79.7
  hsa-miR-634 | 79.3 | 71.2
  hsa-miR-4769-3p | 77.5 | 72.9
  hsa-miR-6507-3p | 76.6 | 72.9
  hsa-miR-3907 | 72.1 | 79.7
  hsa-miR-4634 | 73.0 | 78.0
  hsa-miR-563 | 73.9 | 74.6
  hsa-miR-892b | 73.9 | 74.6
  hsa-miR-103a-2-5p | 74.8 | 71.2
  hsa-miR-2392 | 73.9 | 72.9
  hsa-miR-3127-5p | 72.1 | 76.3
  hsa-miR-338-5p | 73.0 | 74.6
  hsa-miR-3614-5p | 73.9 | 72.9
  hsa-miR-4499 | 70.3 | 79.7
  hsa-miR-3667-5p | 74.8 | 69.5
  hsa-miR-1290 | 68.5 | 78.0
  hsa-miR-130b-5p | 75.7 | 62.7
  hsa-miR-4449 | 73.0 | 67.8
  hsa-miR-4695-5p | 70.3 | 67.8
  hsa-miR-4271 | 67.6 | 71.2
  hsa-miR-4651 | 69.4 | 67.8
  hsa-miR-340-5p | 63.1 | 74.6
  hsa-miR-133b | 67.6 | 61.0
  hsa-miR-199b-5p | 70.3 | 55.9
  hsa-miR-200c-3p | 67.6 | 61.0
  hsa-miR-4257 | 63.1 | 69.5
  hsa-miR-150-3p | 62.2 | 69.5
  hsa-miR-30c-1-3p | 68.5 | 57.6
  hsa-miR-139-3p | 64.9 | 62.7
  hsa-miR-625-3p | 62.2 | 67.8
  hsa-miR-106b-3p | 67.6 | 54.2
  hsa-miR-409-3p | 63.1 | 62.7
  hsa-miR-1237-3p | 63.1 | 61.0
  hsa-miR-5571-5p | 66.7 | 54.2
  hsa-miR-652-5p | 63.1 | 61.0
  hsa-miR-196b-5p | 61.3 | 62.7
  hsa-miR-22-5p | 64.9 | 55.9
  hsa-miR-338-3p | 64.0 | 55.9
  hsa-miR-26b-3p | 62.2 | 55.9
  hsa-miR-4261 | 55.9 | 67.8
  hsa-miR-345-5p | 60.4 | 57.6
  hsa-miR-10a-5p | 58.6 | 59.3
  hsa-miR-3176 | 56.8 | 62.7
  hsa-miR-1224-5p | 56.8 | 61.0
  hsa-miR-4462 | 55.9 | 62.7
  hsa-miR-4728-3p | 58.6 | 57.6
  hsa-miR-193a-5p | 59.5 | 54.2
  hsa-miR-664b-5p | 55.9 | 61.0
  hsa-miR-3141 | 53.2 | 64.4
  hsa-miR-6075 | 55.9 | 59.3
  hsa-miR-6086 | 55.0 | 61.0
  hsa-miR-99b-5p | 55.9 | 59.3
  hsa-miR-1307-3p | 58.6 | 52.5
  hsa-miR-148b-5p | 56.8 | 55.9
  hsa-miR-15a-3p | 59.5 | 50.8
  hsa-miR-6513-3p | 61.3 | 47.5
  hsa-miR-590-5p | 54.1 | 57.6
  hsa-miR-199a-3p | 52.3 | 59.3
  hsa-miR-301a-3p | 55.0 | 52.5
  hsa-miR-4698 | 51.4 | 59.3
  hsa-miR-491-5p | 56.8 | 49.2
  hsa-miR-4701-5p | 53.2 | 54.2
  hsa-miR-572 | 53.2 | 54.2
  hsa-let-7e-5p | 52.3 | 54.2
  hsa-miR-134 | 52.3 | 54.2
  hsa-miR-335-5p | 51.4 | 54.2
  hsa-miR-4646-3p | 54.1 | 49.2
  hsa-miR-4463 | 51.4 | 52.5
  hsa-miR-5690 | 56.8 | 39.0
  hsa-miR-1972 | 46.8 | 50.8
  hsa-miR-769-5p | 48.6 | 47.5
  hsa-miR-126-5p | 43.2 | 55.9
  hsa-miR-192-3p | 52.3 | 39.0
  hsa-miR-4800-5p | 42.3 | 52.5
  hsa-miR-212-3p | 42.3 | 50.8
  hsa-miR-5010-3p | 43.2 | 49.2
  hsa-miR-641 | 48.6 | 39.0
  hsa-miR-3648 | 40.5 | 50.8
  hsa-miR-548ai | 45.9 | 40.7
  hsa-miR-3663-3p | 42.3 | 44.1
  hsa-miR-4298 | 38.7 | 49.2
  hsa-miR-4707-3p | 41.4 | 44.1
  hsa-miR-1273e | 38.7 | 47.5
  hsa-miR-487b | 36.9 | 49.2
  hsa-miR-1227-3p | 40.5 | 40.7
  hsa-miR-18a-3p | 43.2 | 35.6
  hsa-miR-769-3p | 40.5 | 39.0
  hsa-miR-598 | 39.6 | 39.0
  hsa-miR-1273f | 38.7 | 37.3
  hsa-miR-663a | 38.7 | 37.3
  hsa-miR-2110 | 36.9 | 39.0
  hsa-miR-371a-5p | 34.2 | 42.4
  hsa-miR-483-3p | 36.0 | 39.0
  hsa-miR-5195-3p | 37.8 | 35.6
  hsa-miR-654-3p | 35.1 | 35.6
  hsa-miR-877-3p | 34.2 | 37.3
  hsa-miR-3190-5p | 34.2 | 35.6
  hsa-miR-4697-5p | 34.2 | 35.6
  hsa-miR-617 | 36.0 | 32.2
  hsa-miR-4324 | 35.1 | 30.5
  hsa-miR-4534 | 31.5 | 35.6
  hsa-miR-4633-5p | 28.8 | 39.0
  hsa-miR-4538 | 27.9 | 39.0
  hsa-miR-664a-5p | 29.7 | 35.6
  hsa-miR-4312 | 26.1 | 37.3
  hsa-miR-6076 | 25.2 | 35.6
  hsa-miR-5585-3p | 28.8 | 27.1
  hsa-miR-125b-1-3p | 25.2 | 32.2
  hsa-miR-4632-5p | 27.0 | 28.8
  hsa-miR-139-5p | 27.9 | 25.4
  hsa-miR-4767 | 33.3 | 15.3
  hsa-miR-34a-5p | 27.9 | 22.0
  hsa-miR-4455 | 25.2 | 27.1
  hsa-miR-330-3p | 28.8 | 18.6
  hsa-miR-1180 | 25.2 | 23.7
  hsa-miR-193b-3p | 28.8 | 16.9
  hsa-miR-4784 | 20.7 | 30.5
  hsa-miR-4667-5p | 23.4 | 23.7
  hsa-miR-660-3p | 23.4 | 23.7
  hsa-miR-4731-3p | 22.5 | 23.7
  hsa-miR-503-5p | 24.3 | 20.3
  hsa-miR-378g | 18.0 | 27.1
  hsa-miR-4481 | 19.8 | 23.7
  hsa-miR-138-2-3p | 18.9 | 23.7
  hsa-miR-1469 | 20.7 | 20.3
  hsa-miR-4327 | 21.6 | 18.6
  hsa-miR-1236-5p | 17.1 | 23.7
  hsa-miR-152 | 18.0 | 22.0
  hsa-miR-21-3p | 18.9 | 20.3
  hsa-miR-4697-3p | 16.2 | 25.4
  hsa-miR-548aa | 17.1 | 23.7
  hsa-miR-636 | 19.8 | 18.6
  hsa-miR-767-3p | 18.0 | 22.0
  hsa-miR-4689 | 23.4 | 8.5
  hsa-miR-3679-3p | 19.8 | 13.6
  hsa-miR-4326 | 15.3 | 22.0
  hsa-miR-2276 | 17.1 | 16.9
  hsa-miR-3137 | 17.1 | 16.9
  hsa-miR-4734 | 16.2 | 18.6
  hsa-miR-181c-5p | 18.0 | 13.6
  hsa-miR-921 | 17.1 | 15.3
  hsa-miR-3688-3p | 15.3 | 16.9
  hsa-miR-4274 | 15.3 | 16.9
  hsa-miR-4758-5p | 16.2 | 13.6
  hsa-miR-5010-5p | 15.3 | 15.3
  hsa-miR-4488 | 13.5 | 16.9
  hsa-miR-483-5p | 14.4 | 15.3
  hsa-miR-542-5p | 15.3 | 13.6
  hsa-miR-623 | 11.7 | 20.3
  hsa-miR-650 | 9.9 | 23.7
  hsa-miR-3188 | 11.7 | 18.6
  hsa-miR-378b | 10.8 | 20.3
  hsa-miR-576-5p | 12.6 | 16.9
  hsa-miR-20a-3p | 15.3 | 10.2
  hsa-miR-4487 | 15.3 | 10.2
  hsa-miR-1976 | 12.6 | 13.6
  hsa-miR-3605-3p | 12.6 | 13.6
  hsa-miR-4647 | 9.9 | 18.6
  hsa-miR-4700-3p | 11.7 | 15.3
  hsa-miR-6503-3p | 12.6 | 13.6
  hsa-miR-3615 | 10.8 | 13.6
  hsa-miR-424-3p | 10.8 | 13.6
  hsa-miR-4636 | 11.7 | 11.9
  hsa-miR-4646-5p | 9.0 | 16.9
  hsa-miR-3610 | 12.6 | 8.5
  hsa-miR-557 | 9.9 | 13.6
  hsa-miR-718 | 14.4 | 5.1
  hsa-miR-193b-5p | 9.0 | 13.6
  hsa-miR-3692-5p | 12.6 | 6.8
  hsa-miR-509-3-5p | 11.7 | 8.5
  hsa-miR-1470 | 10.8 | 8.5
  hsa-miR-28-3p | 8.1 | 13.6
  hsa-miR-378f | 10.8 | 8.5
  hsa-miR-4252 | 6.3 | 16.9
  hsa-miR-4417 | 11.7 | 6.8
  hsa-miR-4498 | 10.8 | 8.5
  hsa-miR-491-3p | 8.1 | 13.6
  hsa-miR-495-3p | 7.2 | 15.3
  hsa-miR-5096 | 12.6 | 5.1
  hsa-miR-1229-3p | 6.3 | 15.3
  hsa-miR-299-5p | 6.3 | 15.3
  hsa-miR-3138 | 6.3 | 15.3
  hsa-miR-335-3p | 8.1 | 11.9
  hsa-miR-3682-3p | 8.1 | 11.9
  hsa-miR-485-3p | 8.1 | 11.9
  hsa-miR-630 | 7.2 | 13.6
  hsa-miR-936 | 9.0 | 10.2
  hsa-miR-101-5p | 10.8 | 5.1
  hsa-miR-122-5p | 9.9 | 6.8
  hsa-miR-4446-3p | 5.4 | 15.3
  hsa-miR-4518 | 8.1 | 10.2
  hsa-miR-4640-3p | 6.3 | 13.6
  hsa-miR-5189 | 8.1 | 10.2
  hsa-miR-6129 | 8.1 | 10.2
  hsa-miR-1471 | 8.1 | 8.5
  hsa-miR-29b-2-5p | 8.1 | 8.5
  hsa-miR-5003-5p | 5.4 | 13.6
  hsa-miR-1273c | 6.3 | 10.2
  hsa-miR-190a | 9.0 | 5.1
  hsa-miR-3675-3p | 8.1 | 6.8
  hsa-miR-6511b-5p | 5.4 | 11.9
  hsa-miR-1291 | 4.5 | 11.9
  hsa-miR-3934-5p | 4.5 | 11.9
  hsa-miR-4737 | 7.2 | 6.8
  hsa-miR-486-3p | 6.3 | 8.5
  hsa-miR-5580-3p | 2.7 | 15.3
  hsa-miR-671-3p | 7.2 | 6.8
  hsa-miR-154-5p | 6.3 | 6.8
  hsa-miR-3158-5p | 7.2 | 5.1
  hsa-miR-337-3p | 3.6 | 11.9
  hsa-miR-363-5p | 4.5 | 10.2
  hsa-miR-376a-3p | 3.6 | 11.9
  hsa-miR-5190 | 3.6 | 11.9
  hsa-miR-5701 | 6.3 | 6.8
  hsa-miR-770-5p | 3.6 | 11.9
  hsa-miR-1226-5p | 3.6 | 10.2
  hsa-miR-1267 | 6.3 | 5.1
  hsa-miR-1306-3p | 6.3 | 5.1
  hsa-miR-3154 | 4.5 | 8.5
  hsa-miR-329 | 3.6 | 10.2
  hsa-miR-4659b-3p | 7.2 | 3.4
  hsa-miR-6134 | 3.6 | 10.2
  hsa-miR-181a-3p | 4.5 | 6.8
  hsa-miR-1827 | 5.4 | 5.1
  hsa-miR-3926 | 2.7 | 10.2
  hsa-miR-662 | 4.5 | 6.8
  hsa-miR-127-3p | 4.5 | 5.1
  hsa-miR-148a-5p | 3.6 | 6.8
  hsa-miR-18b-3p | 3.6 | 6.8
  hsa-miR-202-3p | 2.7 | 8.5
  hsa-miR-4325 | 2.7 | 8.5
  hsa-miR-4673 | 5.4 | 3.4
  hsa-miR-4730 | 6.3 | 1.7
  hsa-miR-489 | 4.5 | 5.1
  hsa-miR-584-3p | 4.5 | 5.1
  hsa-miR-6720-3p | 1.8 | 10.2
  hsa-let-7i-3p | 5.4 | 1.7
  hsa-miR-1307-5p | 3.6 | 5.1
  hsa-miR-204-5p | 4.5 | 3.4
  hsa-miR-218-5p | 4.5 | 3.4
  hsa-miR-378e | 3.6 | 5.1
  hsa-miR-3911 | 2.7 | 6.8
  hsa-miR-543 | 3.6 | 5.1
  hsa-miR-5703 | 3.6 | 5.1
  hsa-miR-589-3p | 3.6 | 5.1
  hsa-miR-885-5p | 1.8 | 8.5
  hsa-let-7g-3p | 3.6 | 3.4
  hsa-miR-1185-2-3p | 4.5 | 1.7
  hsa-miR-1238-5p | 3.6 | 3.4
  hsa-miR-19b-1-5p | 3.6 | 3.4
  hsa-miR-3130-5p | 2.7 | 5.1
  hsa-miR-3163 | 3.6 | 3.4
  hsa-miR-377-3p | 2.7 | 5.1
  hsa-miR-421 | 2.7 | 5.1
  hsa-miR-4419a | 2.7 | 5.1
  hsa-miR-4425 | 3.6 | 3.4
  hsa-miR-4470 | 3.6 | 3.4
  hsa-miR-4539 | 2.7 | 5.1
  hsa-miR-516a-5p | 3.6 | 3.4
  hsa-miR-610 | 4.5 | 1.7
  hsa-miR-628-5p | 3.6 | 3.4
  hsa-miR-99b-3p | 2.7 | 5.1
  hsa-let-7f-2-3p | 2.7 | 3.4
  hsa-miR-193a-3p | 0.9 | 6.8
  hsa-miR-195-3p | 2.7 | 3.4
  hsa-miR-221-5p | 3.6 | 1.7
  hsa-miR-223-5p | 4.5 | 0.0
  hsa-miR-23a-5p | 1.8 | 5.1
  hsa-miR-25-5p | 1.8 | 5.1
  hsa-miR-3616-3p | 0.9 | 6.8
  hsa-miR-376c-3p | 1.8 | 5.1
  hsa-miR-4701-3p | 2.7 | 3.4
  hsa-miR-4743-5p | 1.8 | 5.1
  hsa-miR-5008-5p | 1.8 | 5.1
  hsa-miR-570-3p | 2.7 | 3.4
  hsa-miR-595 | 1.8 | 5.1
  hsa-miR-6716-3p | 3.6 | 1.7
  hsa-miR-887 | 2.7 | 3.4
  hsa-miR-1299 | 0.9 | 5.1
  hsa-miR-133a | 2.7 | 1.7
  hsa-miR-198 | 1.8 | 3.4
  hsa-miR-3622b-5p | 0.9 | 5.1
  hsa-miR-373-5p | 3.6 | 0.0
  hsa-miR-3917 | 0.9 | 5.1
  hsa-miR-409-5p | 1.8 | 3.4
  hsa-miR-4440 | 2.7 | 1.7
  hsa-miR-4514 | 0.9 | 5.1
  hsa-miR-4535 | 0.9 | 5.1
  hsa-miR-4668-5p | 0.9 | 5.1
  hsa-miR-4776-5p | 0.9 | 5.1
  hsa-miR-4793-3p | 2.7 | 1.7
  hsa-miR-542-3p | 0.9 | 5.1
  hsa-miR-548am-5p | 1.8 | 3.4
  hsa-miR-548q | 1.8 | 3.4
  hsa-miR-582-5p | 2.7 | 1.7
  hsa-miR-654-5p | 1.8 | 3.4
  hsa-miR-758-3p | 2.7 | 1.7
  hsa-miR-760 | 0.0 | 6.8
  hsa-miR-765 | 1.8 | 3.4
  hsa-miR-875-5p | 1.8 | 3.4
  hsa-miR-106a-3p | 2.7 | 0.0
  hsa-miR-1236-3p | 0.0 | 5.1
  hsa-miR-1255b-5p | 1.8 | 1.7
  hsa-miR-181c-3p | 2.7 | 0.0
  hsa-miR-26a-2-3p | 0.9 | 3.4
  hsa-miR-298 | 0.9 | 3.4
  hsa-miR-3194-5p | 0.9 | 3.4
  hsa-miR-3620-3p | 1.8 | 1.7
  hsa-miR-374a-3p | 1.8 | 1.7
  hsa-miR-411-3p | 1.8 | 1.7
  hsa-miR-4475 | 0.9 | 3.4
  hsa-miR-4476 | 0.9 | 3.4
  hsa-miR-4716-5p | 1.8 | 1.7
  hsa-miR-4762-3p | 1.8 | 1.7
  hsa-miR-544a | 1.8 | 1.7
  hsa-miR-548d-5p | 1.8 | 1.7
  hsa-miR-561-3p | 1.8 | 1.7
  hsa-miR-5695 | 2.7 | 0.0
  hsa-miR-580 | 1.8 | 1.7
  hsa-miR-612 | 1.8 | 1.7
  hsa-miR-622 | 0.9 | 3.4
  hsa-miR-670 | 1.8 | 1.7
  hsa-miR-744-3p | 1.8 | 1.7
  hsa-let-7a-3p | 0.9 | 1.7
  hsa-miR-1255a | 0.9 | 1.7
  hsa-miR-1270 | 0.9 | 1.7
  hsa-miR-185-3p | 0.0 | 3.4
  hsa-miR-186-3p | 0.0 | 3.4
  hsa-miR-187-5p | 0.9 | 1.7
  hsa-miR-194-3p | 1.8 | 0.0
  hsa-miR-200b-5p | 0.9 | 1.7
  hsa-miR-2052 | 0.0 | 3.4
  hsa-miR-224-5p | 0.9 | 1.7
  hsa-miR-2964a-5p | 0.9 | 1.7
  hsa-miR-29b-1-5p | 0.9 | 1.7
  hsa-miR-30d-3p | 0.0 | 3.4
  hsa-miR-3150b-5p | 1.8 | 0.0
  hsa-miR-3184-3p | 0.9 | 1.7
  hsa-miR-32-3p | 0.9 | 1.7
  hsa-miR-323a-3p | 1.8 | 0.0
  hsa-miR-3663-5p | 1.8 | 0.0
  hsa-miR-370 | 0.9 | 1.7
  hsa-miR-376a-5p | 0.9 | 1.7
  hsa-miR-381-3p | 0.9 | 1.7
  hsa-miR-3924 | 0.0 | 3.4
  hsa-miR-3945 | 0.9 | 1.7
  hsa-miR-422a | 1.8 | 0.0
  hsa-miR-4289 | 0.9 | 1.7
  hsa-miR-432-3p | 0.0 | 3.4
  hsa-miR-4468 | 0.9 | 1.7
  hsa-miR-452-3p | 0.9 | 1.7
  hsa-miR-452-5p | 0.0 | 3.4
  hsa-miR-4714-5p | 0.9 | 1.7
  hsa-miR-504 | 1.8 | 0.0
  hsa-miR-5088 | 0.0 | 3.4
  hsa-miR-518b | 0.9 | 1.7
  hsa-miR-545-3p | 0.9 | 1.7
  hsa-miR-545-5p | 0.9 | 1.7
  hsa-miR-548at-5p | 0.9 | 1.7
  hsa-miR-556-3p | 0.9 | 1.7
  hsa-miR-559 | 0.0 | 3.4
  hsa-miR-5686 | 0.9 | 1.7
  hsa-miR-5692a | 0.0 | 3.4
  hsa-miR-586 | 0.9 | 1.7
  hsa-miR-590-3p | 1.8 | 0.0
  hsa-miR-601 | 0.9 | 1.7
  hsa-miR-607 | 0.9 | 1.7
  hsa-miR-619 | 0.0 | 3.4
  hsa-miR-624-3p | 1.8 | 0.0
  hsa-miR-642a-5p | 0.9 | 1.7
  hsa-miR-645 | 0.9 | 1.7
  hsa-miR-668 | 0.9 | 1.7
  hsa-miR-6722-3p | 1.8 | 0.0
  hsa-miR-675-5p | 0.9 | 1.7
  hsa-miR-888-3p | 0.9 | 1.7
  hsa-miR-937-3p | 0.9 | 1.7
  hsa-miR-939-3p | 0.9 | 1.7
  hsa-miR-10b-3p | 0.0 | 1.7
  hsa-miR-10b-5p | 0.0 | 1.7
  hsa-miR-1183 | 0.0 | 1.7
  hsa-miR-1208 | 0.0 | 1.7
  hsa-miR-1226-3p | 0.0 | 1.7
  hsa-miR-1228-5p | 0.0 | 1.7
  hsa-miR-124-3p | 0.9 | 0.0
  hsa-miR-124-5p | 0.0 | 1.7
  hsa-miR-1247-3p | 0.9 | 0.0
  hsa-miR-1261 | 0.0 | 1.7
  hsa-miR-1269a | 0.0 | 1.7
  hsa-miR-1273d | 0.9 | 0.0
  hsa-miR-1285-5p | 0.0 | 1.7
  hsa-miR-1287 | 0.0 | 1.7
  hsa-miR-1296 | 0.0 | 1.7
  hsa-miR-143-3p | 0.9 | 0.0
  hsa-miR-1538 | 0.0 | 1.7
  hsa-miR-16-1-3p | 0.9 | 0.0
  hsa-miR-184 | 0.9 | 0.0
  hsa-miR-188-3p | 0.9 | 0.0
  hsa-miR-1909-5p | 0.0 | 1.7
  hsa-miR-1910 | 0.0 | 1.7
  hsa-miR-196a-3p | 0.9 | 0.0
  hsa-miR-19a-5p | 0.0 | 1.7
  hsa-miR-19b-2-5p | 0.9 | 0.0
  hsa-miR-205-5p | 0.9 | 0.0
  hsa-miR-206 | 0.0 | 1.7
  hsa-miR-20b-3p | 0.9 | 0.0
  hsa-miR-2115-5p | 0.9 | 0.0
  hsa-miR-218-1-3p | 0.0 | 1.7
  hsa-miR-218-2-3p | 0.9 | 0.0
  hsa-miR-2277-3p | 0.0 | 1.7
  hsa-miR-2681-3p | 0.9 | 0.0
  hsa-miR-26a-1-3p | 0.9 | 0.0
  hsa-miR-27b-5p | 0.0 | 1.7
  hsa-miR-297 | 0.0 | 1.7
  hsa-miR-29a-5p | 0.0 | 1.7
  hsa-miR-300 | 0.9 | 0.0
  hsa-miR-301b | 0.9 | 0.0
  hsa-miR-302b-3p | 0.0 | 1.7
  hsa-miR-30a-3p | 0.9 | 0.0
  hsa-miR-3132 | 0.0 | 1.7
  hsa-miR-3149 | 0.0 | 1.7
  hsa-miR-3157-5p | 0.0 | 1.7
  hsa-miR-3161 | 0.0 | 1.7
  hsa-miR-32-5p | 0.9 | 0.0
  hsa-miR-330-5p | 0.9 | 0.0
  hsa-miR-33a-3p | 0.9 | 0.0
  hsa-miR-33b-5p | 0.0 | 1.7
  hsa-miR-34c-3p | 0.0 | 1.7
  hsa-miR-3591-3p | 0.0 | 1.7
  hsa-miR-3607-3p | 0.9 | 0.0
  hsa-miR-3654 | 0.0 | 1.7
  hsa-miR-3666 | 0.0 | 1.7
  hsa-miR-367-5p | 0.9 | 0.0
  hsa-miR-374b-3p | 0.9 | 0.0
  hsa-miR-379-3p | 0.9 | 0.0
  hsa-miR-380-5p | 0.9 | 0.0
  hsa-miR-3935 | 0.0 | 1.7
  hsa-miR-3937 | 0.0 | 1.7
  hsa-miR-3942-3p | 0.9 | 0.0
  hsa-miR-3976 | 0.0 | 1.7
  hsa-miR-410 | 0.0 | 1.7
  hsa-miR-4259 | 0.0 | 1.7
  hsa-miR-4272 | 0.0 | 1.7
  hsa-miR-4290 | 0.0 | 1.7
  hsa-miR-4294 | 0.0 | 1.7
  hsa-miR-431-5p | 0.0 | 1.7
  hsa-miR-4420 | 0.9 | 0.0
  hsa-miR-4422 | 0.0 | 1.7
  hsa-miR-4489 | 0.0 | 1.7
  hsa-miR-4500 | 0.9 | 0.0
  hsa-miR-450a-5p | 0.9 | 0.0
  hsa-miR-450b-3p | 0.0 | 1.7
  hsa-miR-451b | 0.9 | 0.0
  hsa-miR-4520b-3p | 0.0 | 1.7
  hsa-miR-4639-3p | 0.9 | 0.0
  hsa-miR-4648 | 0.0 | 1.7
  hsa-miR-4657 | 0.0 | 1.7
  hsa-miR-4677-3p | 0.9 | 0.0
  hsa-miR-4677-5p | 0.9 | 0.0
  hsa-miR-4685-3p | 0.9 | 0.0
  hsa-miR-4694-3p | 0.0 | 1.7
  hsa-miR-4695-3p | 0.0 | 1.7
  hsa-miR-4707-5p | 0.0 | 1.7
  hsa-miR-4710 | 0.0 | 1.7
  hsa-miR-4723-3p | 0.9 | 0.0
  hsa-miR-4726-5p | 0.0 | 1.7
  hsa-miR-4733-3p | 0.0 | 1.7
  hsa-miR-4733-5p | 0.9 | 0.0
  hsa-miR-4736 | 0.0 | 1.7
  hsa-miR-4740-5p | 0.0 | 1.7
  hsa-miR-4755-3p | 0.0 | 1.7
  hsa-miR-4762-5p | 0.0 | 1.7
  hsa-miR-4763-5p | 0.0 | 1.7
  hsa-miR-4785 | 0.0 | 1.7
  hsa-miR-4792 | 0.9 | 0.0
  hsa-miR-4800-3p | 0.9 | 0.0
  hsa-miR-493-5p | 0.0 | 1.7
  hsa-miR-5007-3p | 0.9 | 0.0
  hsa-miR-5011-5p | 0.9 | 0.0
  hsa-miR-5087 | 0.0 | 1.7
  hsa-miR-5093 | 0.0 | 1.7
  hsa-miR-513a-3p | 0.0 | 1.7
  hsa-miR-513c-3p | 0.0 | 1.7
  hsa-miR-517c-3p | 0.0 | 1.7
  hsa-miR-518a-5p | 0.0 | 1.7
  hsa-miR-5196-3p | 0.9 | 0.0
  hsa-miR-520c-3p | 0.9 | 0.0
  hsa-miR-541-3p | 0.0 | 1.7
  hsa-miR-548a-3p | 0.9 | 0.0
  hsa-miR-548ap-3p | 0.9 | 0.0
  hsa-miR-548d-3p | 0.9 | 0.0
  hsa-miR-548e | 0.9 | 0.0
  hsa-miR-552 | 0.9 | 0.0
  hsa-miR-558 | 0.0 | 1.7
  hsa-miR-5591-3p | 0.0 | 1.7
  hsa-miR-5681b | 0.9 | 0.0
  hsa-miR-5692b | 0.9 | 0.0
  hsa-miR-5692c | 0.9 | 0.0
  hsa-miR-571 | 0.0 | 1.7
  hsa-miR-588 | 0.9 | 0.0
  hsa-miR-589-5p | 0.9 | 0.0
  hsa-miR-593-3p | 0.9 | 0.0
  hsa-miR-597 | 0.0 | 1.7
  hsa-miR-609 | 0.9 | 0.0
  hsa-miR-615-3p | 0.0 | 1.7
  hsa-miR-615-5p | 0.0 | 1.7
  hsa-miR-616-5p | 0.9 | 0.0
  hsa-miR-618 | 0.0 | 1.7
  hsa-miR-621 | 0.9 | 0.0
  hsa-miR-631 | 0.0 | 1.7
  hsa-miR-633 | 0.0 | 1.7
  hsa-miR-637 | 0.0 | 1.7
  hsa-miR-639 | 0.9 | 0.0
  hsa-miR-642b-5p | 0.9 | 0.0
  hsa-miR-646 | 0.9 | 0.0
  hsa-miR-6509-3p | 0.9 | 0.0
  hsa-miR-651 | 0.9 | 0.0
  hsa-miR-6511a-3p | 0.0 | 1.7
  hsa-miR-657 | 0.9 | 0.0
  hsa-miR-6722-5p | 0.0 | 1.7
  hsa-miR-708-5p | 0.9 | 0.0
  hsa-miR-767-5p | 0.9 | 0.0
  hsa-miR-875-3p | 0.0 | 1.7
  hsa-miR-876-5p | 0.9 | 0.0
  hsa-miR-877-5p | 0.9 | 0.0
  hsa-miR-891a | 0.9 | 0.0
  hsa-miR-920 | 0.9 | 0.0
  hsa-miR-922 | 0.9 | 0.0
  hsa-miR-924 | 0.0 | 1.7
  hsa-miR-92a-2-5p | 0.9 | 0.0
  hsa-miR-935 | 0.9 | 0.0
  hsa-miR-938 | 0.0 | 1.7
  hsa-miR-943 | 0.9 | 0.0
  hsa-miR-423-5p | 100.0 | 100.0

15. Secondary Outcome: Functional Assessment of Cancer Therapy - Hepatobiliary Questionnaire (FACT-Hep) in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: FACT-Hep consists of 27-item FACT-G, and 18-item Hepatobiliary Subscale. FACT-Hep questionnaire uses 5-point Likert rating scale, range '0'-not at all to '4'. FACT-Hep total score ranges from 0 to 180, where highest score represents maximum achievable quality of life. Domains of FACT-G include Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB) and Functional Well-Being (FWB). Hepatobiliary disease specific items include: swelling or cramps, losing weight, gastrointestinal (GI)-related questions, lack of energy, side effects, pain, fatigue, usual activities, jaundice, fevers, itching, taste of food and chills. Eight of the items (pain, back pain, stomach pain/discomfort, lack of energy, fatigue, nausea, weight loss and jaundice) make up FACT-Hepatobiliary Symptom Index (FHSI-8), and are considered to be symptoms specific to hepatobiliary cancer. Table below included mixed effect model estimated average based on all observed values/time points.
Time Frame: Cycle 1 Day 1 pre-dose and before any other clinical assessments, every 4 weeks thereafter while on study, at end of study treatment/withdrawal, and follow-up and at Day 28 after last dose date
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
units on a scale | 123.33 [120.17 to 126.50] | 135.22 [129.17 to 141.27]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Test type: Superiority or Other; p = 0.0006, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -11.89, 95% CI 2-sided [-18.70 to -5.08]

16. Secondary Outcome: Functional Assessment of Cancer Therapy - General (FACT-G) in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: FACT-G is core questionnaire of Functional Assessment of Chronic Illness Therapy (FACIT) measurement system to evaluate QoL in cancer population. FACT-G consisted of 27 questions grouped in 4 domains of general Health-Related QoL (HRQoL): PWB, SWB, EWB and FWB; each ranging from 0 (not at all) to 4 (very much). FACT-G ranged between 0 and 108. Since questions could be reversed coded, as appropriate, before calculating FACT-G, 0 and 108 could be considered worst and best health states. The below table included the model estimated average based on all the observed values/time points. The mixed effect model was used.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
units on a scale | 71.20 [69.00 to 73.41] | 78.81 [74.68 to 82.93]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.0014, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -7.60, 95% CI 2-sided [-12.27 to -2.94]

17. Secondary Outcome: Functional Assessment of Cancer Therapy (FACT)-Hepatobiliary Symptom Index-8 (FHSI-8) in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: The FACT-Hep includes the FACT-G and a hepatobiliary module. The hepatobiliary disease specific items include: swelling or cramps, losing weight, GI related questions, lack of energy, side effects, pain, fatigue, usual activities, jaundice, fevers, itching, taste of food and chills. Eight of the items (pain, back pain, stomach pain/discomfort, lack of energy, fatigue, nausea, weight loss, and jaundice) make up the FHSI-8, and are considered to be symptoms specific to hepatobiliary cancer. FHSI-8 total score ranges from 0 to 32 where "0" is a severely symptomatic participant and the highest score indicates an asymptomatic participant. The below table included the model estimated average based on all the observed values/time points. The mixed effect model was used.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
units on a scale | 23.42 [22.77 to 24.07] | 26.69 [25.35 to 28.03]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p < 0.0001, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -3.27, 95% CI 2-sided [-4.76 to -1.78]

18. Secondary Outcome: Functional Assessment of Cancer Therapy-G (FACT-G) Subscales in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: FACT-G is core questionnaire of Functional Assessment of Chronic Illness Therapy (FACIT) measurement system to evaluate QoL in cancer population. FACT-G consisted of 27 questions grouped in 4 domains of general HRQoL: PWB, SWB, EWB and FWB. Each of the individual subscale, except EWB has 7 items and each integer scored 0 to 4 making a maximum possible score of 28 (range 0 to 28). EWB has 6 items and each integer scored 0 to 4 making a maximum possible score of 24 (range 0 to 24). For all the 4 scales, higher values correspond to better health. The below table included the model estimated average based on all the observed values/time points. The mixed effect model was used.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
units on a scale
  PWB | 19.39 [18.72 to 20.07] | 23.13 [21.76 to 24.50]
  SWB | 18.94 [18.05 to 19.83] | 20.21 [18.66 to 21.77]
  EWB | 17.23 [16.63 to 17.84] | 17.71 [16.54 to 18.89]
  FWB | 15.76 [14.88 to 16.65] | 17.83 [16.19 to 19.47]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Analysis presented above is for FACT-G PWB. Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Test type: Superiority or Other; p < 0.0001, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -3.74, 95% CI 2-sided [-5.26 to -2.21]
Statistical Analysis 2: Comparison: Axitinib vs Placebo; Analysis presented above is for FACT-G SWB. Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Test type: Superiority or Other; p = 0.1642, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-3.07 to 0.52]
Statistical Analysis 3: Comparison: Axitinib vs Placebo; Analysis presented above is for FACT-G EWB. Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Test type: Superiority or Other; p = 0.4759, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.80 to 0.84]
Statistical Analysis 4: Comparison: Axitinib vs Placebo; Analysis presented above is for FACT-G FWB. Analysis based on repeated measures mixed-effects model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate; Test type: Superiority or Other; p = 0.0288, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-3.92 to -0.21]

19. Secondary Outcome: Functional Assessment of Cancer Therapy - Hepatobiliary Cancer Subscale (FACT Hep-CS18) Questionnaire in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: This subscale consists of 18 items rated on a scale from '0' - not at all to '4' - very much regarding how much each item was present in the last 7 days. FACT-Hep-CS18 total score ranges from 0 to 72. The higher score reflects better QoL or fewer symptoms. The 18 items of this scale are associated with hepatocellular carcinoma. The below table included the model estimated average based on all the observed values/time points. The mixed effect model was used.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
units on a scale | 51.78 [50.46 to 53.10] | 56.74 [54.08 to 59.39]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.0011, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -4.96, 95% CI 2-sided [-7.93 to -1.99]

20. Secondary Outcome: Functional Assessment of Cancer Therapy - Hepatobiliary Cancer Trial Outcome Index (FACT Hep-TOI) Questionnaire in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: The trial outcome index is defined to be the sum (PWB+FWB+HepCS), making it 32 items altogether. Each ranges from '0' - not at all to '4' - very much regarding how much each item was present in the last 7 days. FACT Hep -TOI total score ranges from 0 to 128, where the highest score represents a maximum achievable quality of life. The below table included the model estimated average based on all the observed values/time points. The mixed effect model was used.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
units on a scale | 87.28 [84.98 to 89.58] | 97.73 [93.24 to 102.23]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p < 0.0001, Longitudinal mixed effect analysis — No adjustment made for multiple comparisons; Mean Difference (Final Values) = -10.45, 95% CI 2-sided [-15.49 to -5.42]

21. Secondary Outcome: Time to Deterioration (TTD) Based on the Composite Endpoint in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: TTD analysis was performed for FHSI-8. Time to deterioration was defined as the time between date of randomization and date of the event.
Time Frame: From randomization to death or tumor progression or FHSI-8 mean score decrease >=3 points, whichever comes first
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
months | 1.9 [1.8 to 1.9] | 1.9 [1.8 to 2.7]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Test type: Superiority or Other; p = 0.9182, 1-sided, unstratified log-rank test — The p-value is from a 1-sided log-rank test; Hazard Ratio (HR) = 1.252, 95% CI 2-sided [0.923 to 1.698] — Assuming proportional hazards, a hazard ratio <1 indicates reduction in hazard rate to favor Axitinib, hazard ratio >1 indicates reduction to favor Placebo

22. Secondary Outcome: EuroQoL (EQ-5D)- Health State Profile Utility Score in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. The below table included the model estimated average based on all the observed values/time points. The mixed effect model was used.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
units on a scale | 0.67 [0.63 to 0.70] | 0.79 [0.72 to 0.86]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.0024, Longitudinal mixed effect analysis; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.20 to -0.04]

23. Secondary Outcome: EuroQoL Visual Analogue Scale (EQ-VAS) in Randomized Portion: Overall Between-Treatment Comparison Based on the Repeated Measures Mixed Effects Model
Description: EQ-5D VAS in rates the participant's overall health status using values from 0 (worst imaginable) to 100 (best imaginable). The below table included the model estimated average based on all the observed values/time points. The mixed effect model was used.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 134 | 68
units on a scale | 68.67 [66.11 to 71.23] | 75.70 [70.40 to 81.00]
Statistical Analysis 1: Comparison: Axitinib vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.0193, Longitudinal mixed effect analysis; Mean Difference (Final Values) = -7.03, 95% CI 2-sided [-12.91 to -1.15]

24. Secondary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) in Non-Randomized Portion
Description: Number of Child-Pugh Class B (score 7) participants with DLT was evaluated during Cycle 1 of treatment in the non-randomized portion of the study.
Time Frame: Cycle 1 (4 weeks)
Population: Participants with Child-Pugh Class B, score 7 are only included in this analysis.
Measure: Number; unit: participants
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 0 | 7
participants |  | 2

25. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) in Non-Randomized Portion
Description: An AE was an untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes: death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. The grade of an AE was determined according to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
Time Frame: Up to 28 days after last dose of study drug (up to 6 years)
Population: The safety analysis population included participants who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received.
Measure: Number; unit: participants
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 15 | 7
participants
  Participants with AEs | 15 | 7
  Participants with SAEs | 10 | 3
  Participants >=Grade 3 AEs | 13 | 5
  Participants Grade 5 AEs | 4 | 1

26. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) in Non-Randomized Portion
Description: Treatment-related AE was any untoward medical occurrence in a participant with causal relationship to the study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The grade of an AE was determined according to CTCAE Version 3.0.
Time Frame: Up to 28 days after last dose of study drug (up to 6 years)
Population: as for outcome 25
Measure: Number; unit: participants
Arm/Group | Child-Pugh Class A | Child-Pugh Class B
Number analyzed (Participants) | 15 | 7
participants
  Participants with AEs | 14 (3.55) [94.67 to 237.68] | 6 (2.42) [47.70 to 138.08]
  Participants with SAEs | 2 | 2
  Participants ≥Grade 3 AEs | 9 | 4
  Participants Grade 5 AEs | 0 | 0

27. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) in Randomized Portion
Description: An AE was an untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes: death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. The grade of an AE was determined according to CTCAE Version 3.0.
Time Frame: Up to 28 days after last dose of study drug (up to 6 years)
Population: The safety analysis population included all randomized participants who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received.
Measure: Number; unit: participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 133 | 68
participants
  Participants with AEs | 131 | 63
  Participants with SAEs | 62 | 16
  Participants with Grade >=3 AEs | 109 | 26
  Participants with Grade 5 AEs | 16 | 8

28. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) in Randomized Portion
Description: as for outcome 26
Time Frame: Up to 28 days after last dose of study drug (up to 6 years)
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 133 | 68
participants
  Participants with AEs | 128 | 40
  Participants with SAEs | 24 | 1
  Participants with Grade >=3 AEs | 90 | 12
  Participants with Grade 5 AEs | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up visit (up to 6 years)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- Child-Pugh Class B: Participants with Child-Pugh Class B disease (score 7) at selected sites were initially enrolled only into the non randomized portion of this study to determine the recommended starting dose of axitinib for this population.
Arm/Group | Child-Pugh Class A | Child-Pugh Class B | Axitinib | Placebo
Serious Adverse Events (participants affected / at risk) | 10/15 | 3/7 | 62/133 | 16/68
Other Adverse Events (participants affected / at risk) | 15/15 | 7/7 | 130/133 | 55/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Child-Pugh Class A (N=15) | Child-Pugh Class B (N=7) | Axitinib (N=133) | Placebo (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 3 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 7 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 4 | 0
Disease progression (General disorders) | 3 | 0 | 8 | 4
General physical health deterioration (General disorders) | 0 | 0 | 3 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 4 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abscess rupture (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Ovarian abscess (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Coma hepatic (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 4 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Quadriparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysthymic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Child-Pugh Class A (N=15) | Child-Pugh Class B (N=7) | Axitinib (N=133) | Placebo (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 4 | 0 | 33 | 0
Ocular surface disease (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 5 | 7
Abdominal pain (Gastrointestinal disorders) | 6 | 1 | 45 | 12
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 17 | 3
Anal inflammation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 2 | 21 | 8
Diarrhoea (Gastrointestinal disorders) | 9 | 1 | 71 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 10 | 6
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 35 | 7
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 19 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 26 | 7
Asthenia (General disorders) | 0 | 2 | 27 | 3
Chest discomfort (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Face oedema (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 12 | 2 | 46 | 18
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 2 | 13 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 8 | 0
Oedema (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 4 | 1 | 14 | 10
Pain (General disorders) | 5 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 16 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 9 | 8
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 8 | 2
Alpha 1 foetoprotein increased (Investigations) | 1 | 0 | 0 | 0
Ammonia increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 10 | 4
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 7 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 9 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 5 | 3 | 36 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 5 | 62 | 14
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 9 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 9 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 2 | 8 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3 | 8 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 7 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 11 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 8 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 7 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 9 | 0
Dizziness (Nervous system disorders) | 6 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 21 | 3
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 12 | 3
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 4 | 1 | 27 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 16 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 33 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 13 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 10 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 7
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 2 | 45 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 11 | 8
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 23 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 7 | 3 | 72 | 9
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.